CLINICAL TRIAL: NCT03310281
Title: A Randomized, Double-blind, Controlled, 6-week Trial to Assess the Impact of Novel Digital Interventions Designed to Improve Cognitive Dysfunction as Adjunct Therapy to Antidepressant Medication in Adults With Major Depressive Disorder
Brief Title: Software Treatments for Actively Reducing Severity of Cognitive Deficits in MDD (STARS-MDD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akili Interactive Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Akili-035
Record Dates: First submitted 2017-10-11; First posted 2017-10-16 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Major Depressive Disorder
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALK-T03 (Active Comparator): AKL-T03 is a digital intervention that requires the subject to navigate a character through a game-like space, while collecting objects, in a fixed period of time.
  Interventions: Device: HOLD: Videogame
- AKL-T09 (Active Comparator): AKL-T09 is a digital intervention that requires the subject to spell as many words as possible, by connecting letters in a game-like grid, in a fixed period of time.
  Interventions: Device: HOLD: Videogame

INTERVENTIONS:
Device: HOLD: Videogame — Videogame-like digital therapy

SUMMARY:
The purpose of this study is to evaluate the effects of videogame-like digital therapies as adjunct therapy to antidepressant medications on cognitive deficits associated with major depressive disorder.

DETAILED DESCRIPTION:
The study will be a randomized, parallel group, controlled trial of two videogame-like (iPad-based) digital therapies. The study will consist of 3 primary phases: Pre-screening, Baseline, and Treatment. During the Pre-screening Phase (Day -28 to Day 0), participants will undergo pre-screening to evaluate eligibility for the study. Pre-screening may take place up to 28 days before the Baseline Visit (Day 0). Pre-screening may take place either over the phone, or in the clinic. On Day 0, the Baseline visit will occur wherein additional eligibility criteria will be established. The Treatment Phase (Day 1 to Day 42) will involve using the digital therapy at home for each participant followed by an In-Clinic assessment on Day 42 to assess key outcomes. During the Treatment Phase participants will be instructed to play their videogame-like intervention for approximately 25 minutes per day for 5 days per week. Compliance with treatment/use requirements will be monitored remotely during this phase.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of recurrent Major Depressive Disorder (MDD) according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) as confirmed by MINI Version 7.0.2.
* Pre-Screening (Day≤-28) Remote or In-Clinic
* Screening/Day 0 (in-clinic) including:
* HAM-D-17 score
* BAC Symbol Coding T-test score
* On stable antidepressant medication for ≥8 weeks prior to screening/baseline, with stable dose for ≥4 weeks prior to baseline/baseline, with or without stable adjunct psychotherapy (excluding DBT or CBT) for ≥12 weeks.
* Access to and self-report of ability to connect wireless devices to a functional wireless network
* Ability to follow written and verbal instructions (English) as assessed by the PI and/or study coordinator
* Normal color vision as tested by Ishihara Color Blindness Test
* Able to comply with all testing and requirements

Exclusion Criteria:

* Current controlled (requiring a restricted medication) or uncontrolled, comorbid psychiatric diagnosis with significant symptoms including but not limited to post-traumatic stress disorder, psychosis, bipolar illness, pervasive developmental disorder, severe obsessive compulsive disorder, severe depressive or anxiety disorder, conduct disorder, ADHD or other symptomatic manifestations that in the opinion of the Investigator may confound study data/assessments.
* Initiation or completion of psychotherapy within the last 12 weeks prior to screening/baseline. The participant should inform the Investigator if they intend to change their psychotherapy during the 6 weeks of the study. Participants who have been in psychotherapy consistently for more than 12 weeks may participate if their routine is stable throughout the study.
* Participant is currently considered at risk for attempting suicide by the Investigator, has made a suicide attempt within the past year, or is currently demonstrating active suicidal ideation or self-injurious behavior, as measured by CSSRS.
* Motor condition (e.g. physical deformity of the hands/arms) that prevents game playing as reported by the participant or observed by the Investigator.
* Recent history (6 months prior to screening/baseline) of substance use disorder
* History of seizures (excluding febrile seizures), a tic disorder, significant tics, a current diagnosis of Tourette's Disorder.
* Self-report of recent episodes (within the past week) of nausea, vomiting and/or dizziness.
* Participation in a clinical trial within 3 months prior to screening.
* Color blindness as detected by Ishihara Color Blindness Test
* Regular use of psychoactive drugs other than antidepressants, including stimulants that in the opinion of the Investigator may confound study data/assessments.
* Use of benzodiazepines >3 times per week and/or within 24 hours of baseline and exit visit assessments prohibited.
* Use of marijuana or alcohol on the day of clinical visits before baseline or exit assessments, no tobacco within 30 minutes of TOVA
* Any other medical condition that in the opinion of the Investigator may confound study data/assessments.
* Previous exposure to Akili products.
* Another household member who is/has participated in this trial

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2018-11-14 (Actual)

PRIMARY OUTCOMES:
Change in reaction time to rare target stimuli, from the Test of Variables of Attention (TOVA) | Study Day 0 to Study Day 42
  Compare scores from the first half of the TOVA measured at DAY0/baseline with scores from the first half of the TOVA measured at DAY42/exit between the two treatment groups.

SECONDARY OUTCOMES:
Change in the cognitive component sub-score (items 4-7) of the Cognitive and Physical Functioning Questionnaire (CPFQ) | Study Day 0 to Study Day 42
  Compare cognitive component (items 4-7) of CPFQ scores at DAY0/baseline to (items 4-7) of CPFQ scores at Day42/exit between the two treatment groups
Change in Patient Deficit Questionnaire (PDQ) score | Study Day 0 to Study Day 42
Change in Letter Number Span (LNS) working memory test score | Study Day 0 to Study Day 42
Change in Stroop color and words test score | Study Day 0 to Study Day 42
Change in Trail-making tests A and B scores | Study Day 0 to Study Day 42
Change in BAC Symbol Coding Test score | Study Day 0 to Study Day 42
Change in Trait Adjective Task score | Study Day 0 to Study Day 42

OTHER OUTCOMES:
Exploratory Outcome Measure: Change in Hamilton Depression Scale HAM-D_17 (6 depression-focused subset) | Study Day 0 to Study Day 42
Exploratory Outcome Measure: Change in Patient Health Questionnaire 9 (PHQ-9) score | Study Day 0 to Study Day 42
Exploratory Outcome Measure: Change in Clinical Global Impression Severity and Improvement Scale (CGI-I and CGI-S) scores | Study Day 0 to Study Day 42
Exploratory Outcome Measure: Change in Cognitive and Physical Functioning Questionnaire (CPFQ) total scores | Study Day 0 to Study Day 42
Exploratory Outcome Measure: Change in Patient Deficit Questionnaire (PDQ) score | Study Day 0 to Study Day 42
Exploratory Outcome Measure: Change in Test of Variable of Attention (TOVA) Attention Performance Index (API) | Study Day 0 to Study Day 42
Exploratory Outcome Measure: Change in Quality of Life, Enjoyment and satisfaction Questionnaire - Global Function (Q-LES-Q) scores | Study Day 0 to Study Day 42
Exploratory Outcome Measure: Change in Work & Social Adjustment Scale (WSAS) score | Study Day 0 to Study Day 42
Exploratory Outcome Measure: Change in Emotional Regulation Questionnaire (ERQ) score | Study Day 0 to Study Day 42
Exploratory Outcome Measure: Change in Difficulty in Emotional Regulation Scale (DERS) score | Study Day 0 to Study Day 42

CONTACTS AND LOCATIONS:
Overall Officials: Richard Keefe, PhD, Principal Investigator — Duke Institute for Brain Sciences
Locations (4):
- United States (4):
  - CNS Network, Inc., Garden Grove, California
  - Behavioral Clinical Research, Inc., North Miami, Florida
  - Innovative Clinical Research, Inc., North Miami, Florida
  - Segal Trials, Charleston, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided